CLINICAL TRIAL: NCT01866410
Title: Phase II Trial of XL184 (Cabozantinib) Plus Erlotinib in Patients With Advanced EGFR-Mutant Non-small Cell Lung Cancer (NSCLC) Who Have Progressed on Epidermal Growth Factor Receptor (EGFR) Tyrosine Kinase Inhibitor (TKI) Therapy
Brief Title: Cabozantinib-S-Malate and Erlotinib Hydrochloride in Treating Patients With Previously Treated Metastatic Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01085; NCI-2013-01085 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-125; PHII-125 (Other: City of Hope Comprehensive Cancer Center); 9303 (Other: CTEP); N01CM00038 (NIH); P30CA033572 (NIH)
Record Dates: First submitted 2013-05-28; First posted 2013-05-31 (Estimated); Results first posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-04

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — cabozantinib; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cabozantinib-s-malate, erlotinib hydrochloride) (Experimental): Patients receive cabozantinib-s-malate PO daily and erlotinib hydrochloride PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cabozantinib S-malate; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cabozantinib S-malate — Given PO
  Other Names: BMS-907351; Cabometyx; Cometriq; XL184
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well cabozantinib-s-malate and erlotinib hydrochloride works in treating patients with previously treated metastatic non-small cell lung cancer. Cabozantinib-s-malate and erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Cabozantinib-s-malate may also stop the growth of non-small cell lung cancer by blocking blood flow to the tumor. Giving cabozantinib-s-malate together with erlotinib hydrochloride may be an effective treatment for non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate for efficacy by response rate (RR) when patients with advanced non-small cell lung cancer (NSCLC) harboring an epidermal growth factor receptor (EGFR) mutation who have progressed following EGFR tyrosine kinase inhibitor (TKI) therapy are treated with XL184 (cabozantinib [cabozantinib-s-malate]) and erlotinib (erlotinib hydrochloride).

SECONDARY OBJECTIVES:

I. Determine progression free survival (PFS) for combination XL184 (cabozantinib) and erlotinib in EGFR mutation positive patients following progression on erlotinib.

II. Assess overall survival. III. Evaluate change in tumor growth rate on XL184 (cabozantinib) and erlotinib.

IV. Evaluate type, severity, duration and outcome of toxicities. V. Correlate outcome with tumor biomarkers such as met proto-oncogene (MET) amplification, T790M mutation, and serum markers of the vascular endothelial growth factor (VEGF) and MET pathways in a preliminary manner.

OUTLINE:

Patients receive cabozantinib-s-malate orally (PO) daily and erlotinib hydrochloride PO once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 1 year and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-small cell lung cancer harboring an EGFR mutation; NOTE: EGFR mutational status will be known and assays performed in Clinical Laboratory Improvement Amendments (CLIA) certified laboratories will be accepted
* Patients should have tumor tissue available for retrieval; tissue blocks or unstained slides from the time of original diagnosis are acceptable if repeat biopsy is not indicated
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* Patients must have received prior EGFR TKI therapy for metastatic disease and have documented evidence of radiologic disease progression while on EGFR TKI as treatment immediately prior to enrollment; (patients may have received prior chemotherapy, and retreatment with erlotinib is allowed)
* Eastern Cooperative Oncology Group (ECOG) performance status =< 1 (Karnofsky >= 60%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 × upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3.0 × institutional upper limit of normal
* Lipase < 2.0 x ULN and no radiologic or clinical evidence of pancreatitis
* Creatinine =< 1.5 × ULN OR creatinine clearance >= 50 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Hemoglobin >= 9 g/dL
* Serum albumin >= 2.8 g/dL
* Urine protein/creatinine ratio (UPCR) =< 1
* Serum phosphorus >= lower limit of normal (LLN)
* Calcium >= LLN
* Magnesium >= LLN
* Potassium >= LLN
* Women of childbearing potential must have a negative pregnancy test at screening; women of childbearing potential include women who have experienced menarche and who have not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or are not postmenopausal; postmenopause is defined as amenorrhea >= 12 consecutive months; note: women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antiestrogens, ovarian suppression or any other reversible reason
* Women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of XL184 (cabozantinib) administration; sexually active subjects (men and women) must agree to use medically accepted barrier methods of contraception (e.g., male or female condom) during the course of the study and for 4 months after the last dose of study drug(s), even if oral contraceptives are also used; all subjects of reproductive potential must agree to use both a barrier method and a second method of birth control during the course of the study and for 4 months after the last dose of study drug(s)
* Prior to the first patient registration, this study must have institutional review board (IRB) approval; a copy of the IRB approval for each site involved must be given to the Data Coordinating Center at City of Hope
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* The subject has received cytotoxic chemotherapy (including investigational cytotoxic chemotherapy) or biologic agents (e.g., cytokines or antibodies) within 3 weeks, or nitrosoureas/ mitomycin C within 6 weeks before the first dose of study treatment
* Prior treatment with XL184 (cabozantinib) or other MET/hepatocyte growth factor (HGF) inhibitor
* The subject has received radiation therapy:

  * To the thoracic cavity, abdomen, or pelvis within 2 weeks before the first dose of study treatment, or has ongoing complications, or is without complete recovery and healing from prior radiation therapy
  * To bone or brain metastasis within 14 days before the first dose of study treatment
  * To any other site(s) within 28 days before the first dose of study treatment
* The subject has received prior treatment with a small molecule kinase inhibitor or a hormonal therapy (including investigational kinase inhibitors or hormones) within 14 days or five half-lives of the compound or active metabolites, whichever is longer, before the first dose of study treatment; prior erlotinib is required and does not require a 14-day wash out
* The subject has received any other type of investigational agent within 28 days before the first dose of study treatment
* The subject has not recovered to baseline or Common Terminology Criteria for Adverse Events (CTCAE) =< grade 1 from toxicity due to all prior therapies except alopecia and other non-clinically significant adverse events (AEs)
* The subject has a primary brain tumor
* The subject has active brain metastases or epidural disease; subjects with brain metastases previously treated with whole brain radiation or radiosurgery or subjects with epidural disease previously treated with radiation or surgery who are asymptomatic and do not require steroid treatment for at least 2 weeks before starting study treatment are eligible; baseline brain imaging with contrast-enhanced CT or MRI scans for subjects with known brain metastases is required to confirm eligibility
* The subject has prothrombin time (PT)/ International Normalized Ratio (INR) or partial thromboplastin time (PTT) test >= 1.3 x the laboratory ULN within 14 days before the first dose of study treatment
* The subject requires concomitant treatment, in therapeutic doses, with anticoagulants such as warfarin or warfarin-related agents, heparin, thrombin or Factor Xa inhibitors, or antiplatelet agents (e.g., clopidogrel); low dose aspirin (=< 81 mg/day), low-dose warfarin (=< 1 mg/day), and prophylactic low molecular weight heparin (LMWH) are permitted
* Strong cytochrome P450 (CYP)3A4 inducers and inhibitors should be avoided; selection of alternate concomitant medications with no or minimal CYP3A4 enzyme inhibition potential is recommended; because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx; medical reference texts such as the Physicians' Desk Reference may also provide this information; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* The subject has experienced any of the following:

  * Clinically-significant gastrointestinal bleeding within 6 months before the first dose of study treatment
  * Hemoptysis of >= 0.5 teaspoon (2.5 mL) of red blood within 3 months before the first dose of study treatment
  * Any other signs indicative of pulmonary hemorrhage within 3 months before the first dose of study treatment
* Patients with active bleeding or pathologic conditions that carry high risk of bleeding, such as known bleeding disorder or coagulopathy
* The subject has radiographic evidence of cavitating pulmonary lesion(s)
* The subject has tumor in contact with, invading or encasing any major blood vessels
* The subject has evidence of tumor invading the gastrointestinal (GI) tract (esophagus, stomach, small or large bowel, rectum or anus), or any evidence of endotracheal or endobronchial tumor within 28 days before the first dose of cabozantinib
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders including:

    * Congestive heart failure (CHF): New York Heart Association (NYHA) class III (moderate) or class IV (severe) at the time of screening
    * Concurrent uncontrolled hypertension defined as sustained blood pressure (BP) > 140 mm Hg systolic, or > 90 mm Hg diastolic despite optimal antihypertensive treatment within 7 days of the first dose of study treatment
    * Any history of congenital long QT syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Unstable angina pectoris
      * Clinically-significant cardiac arrhythmias
      * Stroke (including transient ischemic attack [TIA], or other ischemic event)
      * Myocardial infarction
      * Thromboembolic event requiring therapeutic anticoagulation (Note: subjects with a venous filter [e.g. vena cava filter] are not eligible for this study)
  * Gastrointestinal disorders particularly those associated with a high risk of perforation or fistula formation including:

    * Any of the following within 28 days before the first dose of study treatment

      * Intra-abdominal tumor/metastases invading GI mucosa
      * Active peptic ulcer disease
      * Inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis
      * Malabsorption syndrome
    * Any of the following within 6 months before the first dose of study treatment:

      * Abdominal fistula
      * Gastrointestinal perforation
      * Bowel obstruction or gastric outlet obstruction
      * Intra-abdominal abscess; note: Complete resolution of an intra-abdominal abscess must be confirmed prior to initiating treatment with cabozantinib even if the abscess occurred more than 6 months before the first dose of study treatment
  * Other disorders associated with a high risk of fistula formation including percutaneous endoscopic gastrostomy (PEG) tube placement within 3 months before the first dose of study therapy
  * Other clinically significant disorders such as:

    * Active infection requiring systemic treatment within 28 days before the first dose of study treatment
    * Serious non-healing wound/ulcer/bone fracture within 28 days before the first dose of study treatment
    * History of organ transplant
    * Concurrent uncompensated hypothyroidism or thyroid dysfunction within 14 days before the first dose of study treatment
    * History of major surgery as follows:

      * Major surgery within 8 weeks of the first dose of cabozantinib, with complete wound healing; (patients with ongoing wound healing or other complications will be excluded)
      * Minor surgery within 4 weeks of the first dose of cabozantinib; Pleurx catheter placement within 7 days of the first dose of cabozantinib
* The subject is unable to swallow tablets
* The subject has a corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms within 28 days before treatment; note: if initial QTcF is found to be > 500 ms, two additional electrocardiograms (EKGs) separated by at least 3 minutes should be performed; if the average of these three consecutive results for QTcF is =< 500 ms, the subject meets eligibility in this regard
* The subject is unable or unwilling to abide by the study protocol or cooperate fully with the investigator or designee
* The subject has had evidence within 2 years of the start of study treatment of another malignancy which required systemic treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to XL184 (cabozantinib) or erlotinib
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with XL184 (cabozantinib); these potential risks may also apply to other agents used in this study
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-05-20 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Reckamp, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - City of Hope South Pasadena, South Pasadena, California
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania

REFERENCES:
- [Derived] Reckamp KL, Frankel PH, Ruel N, Mack PC, Gitlitz BJ, Li T, Koczywas M, Gadgeel SM, Cristea MC, Belani CP, Newman EM, Gandara DR, Lara PN Jr. Phase II Trial of Cabozantinib Plus Erlotinib in Patients With Advanced Epidermal Growth Factor Receptor (EGFR)-Mutant Non-small Cell Lung Cancer With Progressive Disease on Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor Therapy: A California Cancer Consortium Phase II Trial (NCI 9303). Front Oncol. 2019 Mar 11;9:132. doi: 10.3389/fonc.2019.00132. eCollection 2019. PMID 30915273

RESULTS

PARTICIPANT FLOW:
Groups:
- Cabozantinib-s-malate, Erlotinib Hydrochloride: Patients will receive (A) XL184 (cabozantinib) at 40-mg p.o. daily plus erlotinib at 150-mg p.o. daily in 4-week cycles. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Cabozantinib S-malate: Given PO
  Erlotinib Hydrochloride: Given PO
Period: Overall Study
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride
Started | 37
Completed | 37
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 64 [40 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10
  Black | 1
  Caucasian (non-Hispanic) | 21
  Hispanic/Latino | 4
  Pacific Islander | 1
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride
Number analyzed (Participants) | 37
percentage of participants | 10.8 [0.3 to 21.3]

2. Secondary Outcome: Percentage of Patients With a Greater Than 30% Increase in Tumor Doubling Time
Description: Tumor doubling time was estimated using an exponential growth model. Specifically, the pre-progression scan, and the baseline scan were used to estimate the doubling time prior to enrollment, td = log(2)∗1time/1log(tumor size) [derivation, S(t) = S(to)∗2∧[(t-to)/td] for a parameterization of exponential growth with a doubling time of td. Taking the logarithm on both sides: log(S(t))-log(S(to)) = log(2)∗(t - to)/td or td = log(2)∗(t - to)/[log(S(t))-log(S(to))] = log(2)∗1time/1log(S)], the baseline scan and first evaluation scan were used to determine the doubling time. Based on pre-planned protocol assessment, we estimated the percent of patients that experienced a slowing of tumor kinetics (a 30% increase in the length of time for tumor doubling) based on RECIST v1.1 measurements. Patients who did not get a scan on study, and patients whose pre-progression scans were missing or whose pre-progression tumor size was zero or whose tumor was decreasing prior to enrollment were excluded.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride
Number analyzed (Participants) | 34
percentage of participants | 79 [62 to 91]

3. Secondary Outcome: Number of Adverse Events
Description: Grade 3 & 4 adverse events attributed to treatment agents. Events are graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride
Number analyzed (Participants) | 37
Participants
  Alanine aminotransferase increased | 1
  Aspartate aminotransferase increased | 1
  Dehydration | 2
  Diarrhea | 12
  Fatigue | 2
  Hypertension | 1
  Hypokalemia | 1
  Hypotension | 1
  Lipase increased | 4
  Lymphocyte count decreased | 1
  Myalgia | 1
  Nausea/Vomiting | 3
  Neutrophil count decreased | 1
  Rash acneiform | 2
  Rash maculo-papular | 2
  Serum amylase increased | 4
  Thromboembolic event | 1
  White blood cell decreased | 1

4. Secondary Outcome: Best Response Patient Count
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD), ≥ 20% increase in the sum of the longest diameter of target lesions compared with the smallest-sum longest diameter recorded or the appearance of one or more new lesions; Stable Disease (SD), Neither CR, PR or PD.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride
Number analyzed (Participants) | 37
Participants
  Partial Response | 4
  Stable Disease | 21
  Progressive Disease | 12

5. Secondary Outcome: Progression-free Survival
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Until disease progression or death from any cause, up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride
Number analyzed (Participants) | 37
months | 3.6 [2.0 to 5.6]

6. Secondary Outcome: Overall Survival
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until death from any cause, up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride
Number analyzed (Participants) | 37
months | 13.3 [7.1 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

7. Other Pre Specified Outcome: Progression-free Survival by T790M Mutation Status
Description: Estimated using the product-limit method of Kaplan and Meier. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. DNA was analyzed for the presence of the T790M point mutation.
Time Frame: Until disease progression or death from any cause, up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Positive: Patients will receive (A) XL184 (cabozantinib) at 40-mg p.o. daily plus erlotinib at 150-mg p.o. daily in 4-week cycles. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients had positive T790M status in tissue\blood.
  Cabozantinib S-malate: Given PO
  Erlotinib Hydrochloride: Given PO
- Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Negative: Patients will receive (A) XL184 (cabozantinib) at 40-mg p.o. daily plus erlotinib at 150-mg p.o. daily in 4-week cycles. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients had negative T790M status in tissue\blood.
  Cabozantinib S-malate: Given PO
  Erlotinib Hydrochloride: Given PO
- Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Unknown: Patients will receive (A) XL184 (cabozantinib) at 40-mg p.o. daily plus erlotinib at 150-mg p.o. daily in 4-week cycles. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients had unknown T790M status in tissue\blood.
  Cabozantinib S-malate: Given PO
  Erlotinib Hydrochloride: Given PO
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Positive | Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Negative | Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Unknown
Number analyzed (Participants) | 18 | 13 | 6
months | 2.3 [1.7 to 3.6] | 5.6 [2.8 to 7.3] | 2.4 [1.2 to 12.7]
Statistical Analysis 1: Comparison: Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Positive vs Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Negative vs Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Unknown; Test type: Other; p = 0.4, Log Rank

8. Other Pre Specified Outcome: Overall Survival by T790M Mutation Status
Description: Estimated using the product-limit method of Kaplan and Meier.
Time Frame: Until death from any cause, up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Positive | Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Negative | Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Unknown
Number analyzed (Participants) | 18 | 13 | 6
months | 11.3 [5.6 to NA] — The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment. | 21.2 [5.9 to 21.2] | NA [5.2 to NA] — The upper limit of the 95% confidence interval and median was not calculable because an insufficient number of participants reached the event at the final time point for assessment.
Statistical Analysis 1: Comparison: Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Positive vs Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Negative vs Cabozantinib-s-malate, Erlotinib Hydrochloride, T790M Unknown; Test type: Other; p = 0.5, Log Rank

9. Other Pre Specified Outcome: Changes in VEGF Levels
Time Frame: Baseline up to 6 months after last study treatment
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Changes in HGF Levels
Time Frame: Baseline up to 6 months after last study treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events were recorded and graded throughout the study and until 30 days following the last dose of treatment agent.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Cabozantinib-s-malate, Erlotinib Hydrochloride
All-Cause Mortality (participants affected / at risk) | 32/37
Serious Adverse Events (participants affected / at risk) | 25/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib-s-malate, Erlotinib Hydrochloride (N=37)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 9 (10)
Nausea (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2)
Death NOS (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
bile duct obstruction (Hepatobiliary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Lipase increased (Investigations) | 4 (5)
Lymphocyte count decreased (Investigations) | 2 (3)
Serum amylase increased (Investigations) | 4 (7)
White blood cell decreased (Investigations) | 1 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vasovagal reaction (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib-s-malate, Erlotinib Hydrochloride (N=37)
Anemia (Blood and lymphatic system disorders) | 20 (52)
Palpitations (Cardiac disorders) | 1 (3)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 2 (3)
Hypothyroidism (Endocrine disorders) | 2 (10)
Low testosterone (Endocrine disorders) | 1 (2)
Blurred vision (Eye disorders) | 2 (3)
Dry eye (Eye disorders) | 1 (1)
Glaucoma (Eye disorders) | 1 (8)
bilateral blepharitis (Eye disorders) | 1 (1)
blepharitis (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 11 (23)
Anal pain (Gastrointestinal disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (6)
Burping (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 12 (26)
Diarrhea (Gastrointestinal disorders) | 33 (132)
Dry mouth (Gastrointestinal disorders) | 6 (13)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Dysphagia (Gastrointestinal disorders) | 3 (4)
Flatulence (Gastrointestinal disorders) | 5 (8)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 (6)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 4 (8)
Increased appetite (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 6 (14)
Nausea (Gastrointestinal disorders) | 15 (32)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 3 (3)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (14)
broken tooth (Gastrointestinal disorders) | 1 (2)
Chest tightness (General disorders) | 1 (2)
Chills (General disorders) | 2 (3)
Edema limbs (General disorders) | 6 (9)
Fatigue (General disorders) | 30 (98)
Flu like symptoms (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 10 (16)
Pain (General disorders) | 2 (7)
Swellign in limbs (General disorders) | 1 (1)
body aches (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1)
Fungal & Skin infection (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Papulopustular rash (Infections and infestations) | 2 (3)
Paronychia (Infections and infestations) | 6 (15)
Pharyngitis (Infections and infestations) | 1 (2)
Sinusitis (Infections and infestations) | 1 (3)
Skin infection (Infections and infestations) | 5 (8)
Upper respiratory infection (Infections and infestations) | 3 (5)
Urinary tract infection (Infections and infestations) | 6 (10)
Bruising (Injury, poisoning and procedural complications) | 1 (3)
Activated partial thromboplastin time pr (Investigations) | 1 (2)
Alanine aminotransferase increased (Investigations) | 21 (64)
Alkaline phosphatase increased (Investigations) | 11 (19)
Aspartate aminotransferase increased (Investigations) | 24 (85)
Blood bilirubin increased (Investigations) | 13 (24)
CD4 lymphocytes decreased (Investigations) | 1 (1)
Cardiac troponin I increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 2 (10)
Creatinine increased (Investigations) | 3 (4)
Electrocardiogram QT corrected interval (Investigations) | 1 (1)
GGT increase (Investigations) | 1 (1)
GGT increased (Investigations) | 10 (27)
Hemoglobin increased (Investigations) | 1 (1)
INR increased (Investigations) | 1 (1)
LDH Increase (Investigations) | 2 (2)
LDH Increased (Investigations) | 1 (1)
LDH increase (Investigations) | 1 (1)
LDH increased (Investigations) | 3 (4)
Lipase increased (Investigations) | 10 (17)
Lymphocyte count decreased (Investigations) | 15 (36)
Neutrophil count decreased (Investigations) | 6 (14)
Platelet count decreased (Investigations) | 7 (14)
Serum amylase increased (Investigations) | 16 (46)
Weight gain (Investigations) | 3 (8)
Weight loss (Investigations) | 16 (43)
White blood cell decreased (Investigations) | 11 (43)
blood LDH increase (Investigations) | 6 (9)
blood lactate dehydrogenase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 21 (53)
Dehydration (Metabolism and nutrition disorders) | 4 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 5 (7)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (29)
Hypocalcemia (Metabolism and nutrition disorders) | 14 (27)
Hypoglycemia (Metabolism and nutrition disorders) | 9 (31)
Hypokalemia (Metabolism and nutrition disorders) | 10 (18)
Hypomagnesemia (Metabolism and nutrition disorders) | 8 (14)
Hyponatremia (Metabolism and nutrition disorders) | 12 (33)
Hypophosphatemia (Metabolism and nutrition disorders) | 5 (11)
Obesity (Metabolism and nutrition disorders) | 3 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (6)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (20)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (8)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 5 (7)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 10 (29)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (12)
Aphasia (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (3)
Cold intolerance (Nervous system disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 2 (4)
Dizziness (Nervous system disorders) | 7 (13)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 11 (29)
Headache (Nervous system disorders) | 11 (19)
Lethargy (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 2 (5)
Neuralgia (Nervous system disorders) | 2 (6)
Paresthesia (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (4)
Vasovagal reaction (Nervous system disorders) | 1 (1)
aphasia (Nervous system disorders) | 1 (2)
sensitivity to light and heat (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (10)
Confusion (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 3 (6)
Insomnia (Psychiatric disorders) | 1 (2)
BPH (Renal and urinary disorders) | 1 (2)
Hematuria (Renal and urinary disorders) | 2 (5)
Proteinuria (Renal and urinary disorders) | 7 (9)
URINARY PROBLEMS (Renal and urinary disorders) | 1 (1)
Urinary BPH problem (Renal and urinary disorders) | 1 (3)
Urinary BPH problems (Renal and urinary disorders) | 1 (1)
Urinary Problem BPH (Renal and urinary disorders) | 1 (2)
Urinary Problem PPH (Renal and urinary disorders) | 1 (1)
Urinary Problems BPH (Renal and urinary disorders) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 3 (3)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (43)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 17 (41)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 4 (18)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4 (8)
Runny nose (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Scratchy voice (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 5 (7)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (4)
Callus (Skin and subcutaneous tissue disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cracked nail (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 18 (62)
Facial Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Finger tip/nail cracks (Skin and subcutaneous tissue disorders) | 1 (3)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (2)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (2)
Nail Chenges, NOS (Skin and subcutaneous tissue disorders) | 1 (1)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndro (Skin and subcutaneous tissue disorders) | 3 (7)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 7 (14)
Rash acneiform (Skin and subcutaneous tissue disorders) | 8 (23)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 (59)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (2)
facial rash (Skin and subcutaneous tissue disorders) | 2 (4)
finger tip/nail cracks (Skin and subcutaneous tissue disorders) | 1 (1)
fingertip/nail cracks (Skin and subcutaneous tissue disorders) | 1 (3)
ingrown eyelash (Skin and subcutaneous tissue disorders) | 1 (1)
mild rash (Skin and subcutaneous tissue disorders) | 1 (1)
mild tenderness Callus on foot (Skin and subcutaneous tissue disorders) | 1 (1)
peeling of hands (Skin and subcutaneous tissue disorders) | 1 (2)
rash (Skin and subcutaneous tissue disorders) | 1 (1)
rash erythema (Skin and subcutaneous tissue disorders) | 1 (3)
right hand laceration (Skin and subcutaneous tissue disorders) | 1 (1)
yeast like rash (Skin and subcutaneous tissue disorders) | 1 (2)
yeast-like rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 16 (76)
Hypotension (Vascular disorders) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (1014-01-24): https://cdn.clinicaltrials.gov/large-docs/10/NCT01866410/Prot_SAP_000.pdf